CLINICAL TRIAL: NCT06188208
Title: A Phase 1, Open-Label, 2-Part, Multicenter, First-in-Human Dose Escalation and Dose Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Anti-Tumor Activity of the STAT3 Inhibitor VVD-130850 as Single Agent and in Combination With Checkpoint Inhibition in Participants With Advanced Solid and Hematologic Tumors
Brief Title: A First-in-Human (FIH) Study to Evaluate the Safety and Tolerability of VVD-130850 in Participants With Advanced Solid and Hematologic Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vividion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VVD-130850-01; 2023-508386-32-00 (Other: EU CTIS Number)
Record Dates: First submitted 2023-12-13; First posted 2024-01-03 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumors; Advanced Hematologic Tumors
Keywords: VVD-130850; Phase I; First in Human; Cancer; small molecule; STAT3; NSCLC; STK11; LKB1; immunosuppression; Checkpoint inhibitor; PD-1
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dose Escalation: VVD-130850 Single Agent (Experimental): Participants will receive ascending doses of VVD-130850, orally, once daily in 21-day treatment cycles during the dose escalation phase.
  Interventions: Drug: VVD-130850
- Dose Escalation: VVD-130850 + Pembrolizumab Combination Therapy (Experimental): Participants will receive ascending doses of VVD-130850, orally, once daily, along with pembrolizumab intravenous (IV) infusion, every 3 weeks (Q3W) in 21-day treatment cycles during the dose escalation phase.
  Interventions: Drug: VVD-130850; Drug: Pembrolizumab
- Dose Expansion: VVD-130850 Single Agent (Experimental): Participants will receive VVD-130850 at recommended dose for expansion (RDE), orally, once daily in 21-day treatment cycles during the dose expansion phase.
  Interventions: Drug: VVD-130850
- Dose Expansion: VVD-130850 + Pembrolizumab Combination Therapy (Experimental): Participants will receive VVD-130850 at RDE orally, once daily along with pembrolizumab IV infusion, Q3W in 21-day treatment cycles during the dose expansion phase.
  Interventions: Drug: VVD-130850; Drug: Pembrolizumab

INTERVENTIONS:
Drug: VVD-130850 — Oral tablets
Drug: Pembrolizumab — IV infusion
  Arms: Dose Escalation: VVD-130850 + Pembrolizumab Combination Therapy; Dose Expansion: VVD-130850 + Pembrolizumab Combination Therapy

SUMMARY:
A FIH study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of VVD-130850, as single agent and in combination with checkpoint inhibition, in participants with advanced solid and hematologic tumors.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically or cytologically confirmed metastatic or unresectable solid tumor or advanced non-Hodgkin's lymphoma (NHL).
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
3. Adequate organ and bone marrow function as defined in the protocol.
4. For Combination Therapy Expansion:

   * Serine/threonine kinase 11/ liver kinase B1 (STK11/LKB1) mutated non-small cell lung cancer (NSCLC) as assessed by historical (local) test.
   * Must be refractory to or have progressed on or after a platinum-based doublet regimen and an immune checkpoint inhibitor (CPI). These therapies could have been given in the same line of therapy or different lines of therapy.
5. Measurable disease by RECIST version 1.1 as assessed by the Investigator.

Key Exclusion Criteria:

1. Have a diagnosis of immunodeficiency or are receiving systematic steroid therapy or any other form of immunosuppressive therapy.
2. Prior allogeneic transplantation.
3. History of cardiac diseases as defined in detail in the protocol.
4. Clinically significant infection or any eye infection.
5. Active central nervous system (CNS) malignancies (previously treated CNS malignancies are not exclusionary).
6. Combination Therapy Expansion:

   * Known hypersensitivity or contraindication to pembrolizumab or any of its components.
   * Any prior toxicity (Grade 3 or 4) related to immunotherapy leading to treatment discontinuation with the exception of the history of immunotherapy-related endocrinopathy controlled with ongoing medical management (e.g., hypothyroidism, adrenal insufficiency, diabetes).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation: Incidence and Severity of Dose-limiting Toxicities (DLTs) During DLT Observation Period | From Day 1 to Day 21 of Cycle 1 [cycle length=21 days]
  Incidence and severity of DLTs will be assessed per DLT criteria set forth in the protocol based on adverse events (AEs) evaluated per National Cancer Institute (NCI) - Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Dose Expansion: Number of Participants with AEs and Serious Adverse Events (SAEs) | Up to approximately 4 years
Dose Expansion: Number of Participants with Clinically Significant Changes in Vital Signs | Up to approximately 4 years
Dose Expansion: Number of Participants with Clinically Significant Changes in Laboratory Evaluations | Up to approximately 4 years

SECONDARY OUTCOMES:
Dose Escalation: QT/Corrected QT (QTc) Interval and Other Electrocardiogram (ECG) Parameters | Up to approximately 4 years
  Number of participants with changes in QT/QTc interval and other ECG parameters will be assessed.
Dose Escalation: Recommended Dose for Expansion (RDE) of VVD-130850 as a Single Agent and in Combination with Pembrolizumab | Up to approximately 4 years
  The RDE will be based on safety, pharmacokinetics, pharmacodynamic biomarker data, and preliminary anti-tumor activity collected during the study as defined by the safety review committee.
Dose Expansion: Overall Response Rate (ORR) | Up to approximately 4 years
  ORR is defined as the percentage of participants achieving a best overall response of complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator assessment.
Dose Expansion: Duration of Response (DoR) | Up to approximately 4 years
  DOR is defined as the time from initial response of CR or PR to progressive disease or death, whichever comes first per RECIST version 1.1 by investigator assessment.
Dose Expansion: Progression-free Survival (PFS) | Up to approximately 4 years
  PFS is defined as the time from the date of randomization to the time of confirmed disease progression or death, whichever occurs first per RECIST version 1.1 by investigator assessment.
Dose Expansion: Disease Control Rate (DCR) | Up to approximately 4 years
  DCR is defined as the percentage of participants achieving CR or PR, or stable disease (SD) per RECIST version 1.1 by investigator assessment.
Dose Escalation and Expansion: Area Under the Plasma Concentration-time Curve (AUC) of VVD-130850 | Predose and multiple timepoints post-dose from Cycle 1 Day 1 up to Cycle 5 Day 1 (cycle length=21 days)
Dose Escalation and Expansion: Maximum Plasma Concentration (Cmax) of VVD-130850 | Predose and multiple timepoints post-dose from Cycle 1 Day 1 up to Cycle 5 Day 1 (cycle length=21 days)
Dose Escalation and Expansion: Apparent Terminal Half-life (t1/2) of VVD-130850 | Predose and multiple timepoints post-dose from Cycle 1 Day 1 up to Cycle 5 Day 1 (cycle length=21 days)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (9):
  - California Research Institute, Los Angeles, California
  - Florida Cancer Specialists, Sarasota, Florida
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - NEXT Austin, Austin, Texas
  - MDACC, Houston, Texas
  - NEXT Dallas, Irving, Texas
  - NEXT San Antonio, San Antonio, Texas
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
  - NEXT Virginia, Fairfax, Virginia
- Australia (5):
  - Blacktown Hospital, Blacktown, New South Wales
  - Orange Health Service, Orange, New South Wales
  - Gold Coast University Hospital, Southport, Queensland
  - Cancer Research South Australia, Adelaide
  - ICON Cancer Research, South Brisbane
- Spain (6):
  - START Barcelona Hospital HM Nou Delfos, Barcelona
  - Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - NEXT Madrid, Madrid
  - START Madrid CIOCC, Madrid
  - Start Madrid-FJD, Hospital Fundacion Jimenez Diaz, Madrid

IPD SHARING:
Plan to Share IPD: No